CLINICAL TRIAL: NCT06190652
Title: Real-world Experience of Immunotherapy Plus Chemotherapy as First-line Treatment With or Without Radiotherapy for Patients With Advanced Oesophageal Squamous Cell Carcinoma in China
Brief Title: Real-world Experience of ICIs Plus Chemotherapy With or Without Radiotherapy for Advanced ESCC.
Acronym: REICRAE
Status: Completed | Type: Observational
Sponsor: Tianjin Medical University Cancer Institute and Hospital (Other)
Collaborators: Sichuan Cancer Hospital and Research Institute (Other); Henan Cancer Hospital (Other Government); Shanxi Province Cancer Hospital (Other); Hunan Cancer Hospital (Other); The First Affiliated Hospital with Nanjing Medical University (Other); Hebei Medical University Fourth Hospital (Other)
Responsible Party: Sponsor
Other Study IDs: bc2023043
Record Dates: First submitted 2023-12-19; First posted 2024-01-05 (Actual); Last update posted 2024-02-05 (Actual); Status verified 2023-12

CONDITIONS: Metastatic Esophageal Squamous Cell Carcinoma
MeSH Terms: conditions — Esophageal Squamous Cell Carcinoma | interventions — Immunotherapy; Radiotherapy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Arm A: Chemotherapy combined with immunotherapy group
  Interventions: Drug: Chemotherapy combined with immunotherapy
- Arm B: Chemotherapy combined with immunotherapy + radiotherapy group
  Interventions: Drug: Chemotherapy combined with immunotherapy; Radiation: radiotherapy

INTERVENTIONS:
Drug: Chemotherapy combined with immunotherapy — chemotherapy：paclitaxel+platinum-based anticancer drugs immunotherapy：anti-PD-1 Immune checkpoint inhibitors
Radiation: radiotherapy — Intensity-modulated radiation therapy
  Groups: Arm B

SUMMARY:
This study is a multi-center, non-interventional study. Clinicopathologic, treatment , outcome and efficacy data will be collected from medical records in metastatic esophageal squamous cell carcinoma (ESCC) patients.

DETAILED DESCRIPTION:
This study is a multi-center, non-interventional study. Patients' background, treatment pattern, treatment outcome, efficacy will be collected in metastatic esophageal squamous cell carcinoma (ESCC) patients who were treated with chemotherapy combined with immunotherapy as 1st line treatment at approximately 5 institutions. The patients should have received at least 1 cycle of immunotherapy and chemotherapy with or without radiotherapy. Based on these data, overall survival (OS), progression free survival (PFS) from start of 1st line treatment and the role and efficacy of radiotherapy for these patients will be assessed.

ELIGIBILITY:
Inclusion Criteria:

1. Pathologically diagnosed as esophageal squamous cell carcinoma;
2. The clinical stage is IVb stage, that is, non-regional lymph node metastasis and distant organ metastasis (AJCC8th) of esophageal carcinoma.
3. Patients had received no previous systemic therapy
4. Patients who had received at least one cycle of first-line chemotherapy combined with immunotherapy, received or did not receive radiotherapy;
5. Complete medical records;
6. ECOG0-2;

Exclusion Criteria:

1. Surgery for esophageal cancer;
2. Esophageal fistulae due to infiltration of the primary tumour.
3. Risk of gastrointestinal bleeding, oesophageal fistula or oesophageal perforation
4. Those who have a history of autoimmune disease or have been treated with immunosuppressants within the last 3 months.
5. Those who have received organ transplant surgery.
6. Patients with a previous history of malignant tumor (skin basal cell carcinoma and cervical carcinoma in situ) survived tumor-free for 3 years after treatment.

   Except for the above).
7. There are other serious diseases, such as myocardial infarction, cerebral infarction or severe cardiopulmonary insufficiency within 6 months

Ages: 18 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: 1. The clinical stage is IVb stage, that is, non-regional lymph node metastasis and distant organ metastasis (AJCC8th) of esophageal carcinoma.
  2. Patients who had received at least one cycle of first-line chemotherapy combined with immunotherapy, received or did not receive radiotherapy;
  3. Pathologically diagnosed as esophageal squamous cell carcinoma;
Sampling Method: Non-Probability Sample
Enrollment: 728 (Actual)
Dates: Start 2018-10-13 (Actual); Primary Completion 2023-12-04 (Actual); Study Completion 2023-12-04 (Actual)

PRIMARY OUTCOMES:
PFS | up to 2 years
  progression-free survival

SECONDARY OUTCOMES:
OS | up to 2 years
  overall Survival
DoR | up to 2 years
  Duration of ResponseR
ORR | up to 2 years
  Objective Response Rate
RP | up to 2 years
  recurrence recurrence pattern

CONTACTS AND LOCATIONS:
Overall Officials: Wencheng Zhang, M.D., Principal Investigator — Tianjin Medical University Cancer Institute and Hospital
Locations (5):
- China (5):
  - Henan Cancer Hospital, Zhengzhou, Henan
  - Hunan Cancer Hospital, Changsha, Hunan
  - Shanxi Cancer Hospital, Taiyuan, Shanxi
  - Sichuan Cancer Hospital, Chengdu, Sichuan
  - Tianjin Cancer Hospital, Tianjin, Tianjin Municipality

IPD SHARING:
Plan to Share IPD: No